CLINICAL TRIAL: NCT03020485
Title: The Glycaemic Effect of Isomaltulose Consumption in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Melvin Leow, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 2014/01008
Record Dates: First submitted 2017-01-10; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — isomaltulose; Sucrose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isomaltulose (Experimental): 50g of isomaltulose dissolved in 250ml of water
  Interventions: Other: Isomaltulose
- Sucrose (Experimental): 50g of sucrose dissolved in 250ml of water
  Interventions: Other: Sucrose

INTERVENTIONS:
Other: Isomaltulose — Isomaltulose is a disaccharide made up of one molecule glucose and fructose with a (α1-6) linkage.
  Arms: Isomaltulose
Other: Sucrose — Sucrose is normal table sugar
  Arms: Sucrose

SUMMARY:
The objective of this study is to determine the glycaemic effect of isomaltulose and sucrose in Chinese, Indian, Malay, and Caucasian individuals. The current study will provide important information on the potential health benefits of isomaltulose consumption in Asian population. It will also reveal how the three main ethnicities in Singapore respond to isomaltulose and whether the response differs from the Caucasians.

DETAILED DESCRIPTION:
The objective of the present study is to investigate the glycaemic effect of isomaltulose in Chinese, Indians, Malays and Caucasians. This will be a single intervention. Up to fifty participants, consisting of at least ten Chinese, ten Malays, ten Indians, and ten Caucasians completed data sets, aged between 21 and 40 years will be recruited from the general public in Singapore. Participants will be asked to attend two test sessions for this study. Participants will consume either a sucrose drink or an isomaltulose drink (each containing 50 g of available carbohydrate).

ELIGIBILITY:
Inclusion Criteria:

* Chinese, Indian, Malay or Caucasian ethnic origin

Exclusion Criteria:

* People with major chronic disease such as heart disease, cancer or diabetes mellitus
* Individuals with food intolerances or allergies to isomaltulose or sucrose
* Individuals who are taking insulin or drugs known to affect glucose metabolism and body fat distribution
* People with a major medical or surgical event requiring hospitalization within the preceding 3 months
* Individuals with the presence of disease or drugs which influence digestion and absorption of nutrients
* Pregnant women

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in post prandial Blood glucose for 180 minutes period | 180 minutes
  Blood glucose obtained through finger pricks using Hemocue Glucose Analyser

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Leow, MD, Principal Investigator — Clinical Nutrition Research Centre

IPD SHARING:
Plan to Share IPD: No